CLINICAL TRIAL: NCT05602285
Title: IV Dislodgement Device Single Site Comparative Effectiveness Study
Brief Title: IV Dislodgement Comparative Effectiveness Study
Status: Terminated | Type: Observational
Why Stopped: Hospital IV tubing connector did not match Linear health Product connector. Found this out after enrolling 2 patients. Study permanently stopped March 2025 after realizing that our site was not planning to change the IV tubing currently in use
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Sandra Siedlecki, Senior Nurse Scientist, The Cleveland Clinic
Other Study IDs: 22-1051
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: IVF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Usual care group: Usual IV securement
- Dislodgement device group: Usual IV securement plus dislodgement device
  Interventions: Device: Dislodgement device

INTERVENTIONS:
Device: Dislodgement device — Breakaway device that prevents IV dislodgement
  Groups: Dislodgement device group

SUMMARY:
The goal of this comparative effectiveness study is to compare IV dislodgement frequency in medical-surgical patients with continuous IV fluids infusing.

The main question it aims to answer are:

1. To determine if the addition of the break-away IV device within IV tubing and customary IV dressing reduces dislodgment when compared to customary IV dressing alone.

DETAILED DESCRIPTION:
Accidental dislodgement of peripheral venous assess devices occurs in up to 25% of all peripheral IV catheters. Accidental dislodgement is costly in terms of comfort, time, and resources. Dislodged IVs must usually be restarted and during the dislodgement period the patient is not receiving fluids and/or IV medications (delay or missed treatment). A few researchers reported the efficacy of various IV dressings related to their securement capabilities. Although dressings vary, the incidence of dislodgement was not associated with this method. Additionally, researchers have not explored the use of a break-away device that disconnects IV tubing from the IV catheter prior to dislodgement.

The purpose of this study is to determine if the addition of a break-away device results in fewer IV dislodgements than standard care alone. The aims of this study are to determine if the addition of the break-away IV device within IV tubing and customary IV dressing reduces dislodgment when compared to customary IV dressing alone; and to obtain feedback from nurses who used the break-away device regarding its strengths and limitations.

Four similar medical-surgical units at a quaternary care medical center will be used (H80 & 81 and H70 & 71). The floors (70s and 80s) will be randomly assigned to the study or control group by a coin flip at the beginning of the study. Two units will continue with customary IV dressing protocols and two units will use the break-away device in the IV tubing in addition to customary IV dressing.

Unit caregivers will be expected to record an IV dislodgement and restart date on the case report form at the time of the event. A research nurse will round on all patients on each unit daily.

The statistician has determined that to detect a 30% decrease in IV dislodgement, approximately 381 patients per group for 80% power would be required. As attrition is a potential threat for this study an additional 10% will be included in the final sample size calculations. Thus a total sample of 762 patients plus 10% (for attrition) will result in a sample of 838 patients with IVs for this study, to obtain the required 2286 patient days needed for analysis (based on an average of 3 patient days per subject).

For use in the regression model and to adjust (control) for differences in patient or environment characteristics that may impact dislodgement, the investigators will collect the following: patient characteristics (age, race, sex), environmental characteristics (time of day of dislodgment), and IV characteristics (IV catheter size, IV catheter site, right vs left).

ELIGIBILITY:
Inclusion Criteria:

Patient with IV fluids running through peripheral line Adult medical/surgical patients

Exclusion Criteria:

Patients <18 years old Adult patients with central lines (PICC, triple lumen, med-port) No continuous IVF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with IV fluids running through a peripheral line
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of IV dislodgements | 3-day hospital stay
  Frequency of IV dislodgements

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No